CLINICAL TRIAL: NCT07362355
Title: A Multicenter, Randomized, Double-blind, Active-controlled Parallel-group Phase ii Clinical Study to Compare the Efficacy and Safety of SHR4640 Tablets Combined With Febuxostat Tablets at 40 mg/Day Versus Febuxostat Tablets With Dose Escalation in Treatment of Primary Gout and Hyperuricemia Subjects With Inadequate Control on 40 mg/Day Febuxostat
Brief Title: The Efficacy and Safety of SHR4640 Tablet Combined With 40 mg Febuxostat Tablets in the Treatment of Primary Gout and Hyperuricemia
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR4640-204
Record Dates: First submitted 2026-01-15; First posted 2026-01-23 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Primary Gout and Hyperuricemia
MeSH Terms: conditions — Hyperuricemia | interventions — ruzinurad; Febuxostat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Treatment group A (Experimental)
  Interventions: Drug: SHR4640 ；Febuxostat
- Treatment group B (Experimental)
  Interventions: Drug: SHR4640 ; Febuxostat
- Treatment group C (Experimental)
  Interventions: Drug: SHR4640
- Treatment group D (Experimental)
  Interventions: Drug: SHR4640
- Treatment group E (Active Comparator)
  Interventions: Drug: Febuxostat

INTERVENTIONS:
Drug: SHR4640 ；Febuxostat — SHR4640 high dose + Febuxostat
  Arms: Treatment group A
Drug: SHR4640 ; Febuxostat — SHR4640 low dose + Febuxostat
  Arms: Treatment group B
Drug: SHR4640 — SHR4640 high dose
  Arms: Treatment group C
Drug: SHR4640 — SHR4640 low dose
  Arms: Treatment group D
Drug: Febuxostat — Febuxostat
  Arms: Treatment group E

SUMMARY:
SHR4640 tablets is a highly selective and potent URAT1 inhibitors. The study is being conducted to evaluate the efficacy, and safety of SHR4640 tablet combined with 40 mg/d febuxostat tablet in reducing uric acid in subjects with primary gout and hyperuricemia The primary purpose of the study is to evaluate the efficacy and safety of the combination of SHR4640 and 40 mg/d febuxostat compared with 60 mg/d febuxostat in primary gout and hyperuricemia subjects with inadequate control on 40 mg/d febuxostat for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily signed the informed consent, understood the procedures and methods of the study, and was willing to complete the study strictly in accordance with the clinical trial protocol;
2. The screening age should be 18-75 years old (including both ends), male or female;
3. Receive febuxostat at a stable dose of 40 mg/day for ≥6 weeks before randomization; have a fasting serum uric acid level ≥390 µmol/L at the first measurement, and a repeat fasting serum uric acid level ≥360 µmol/L after taking febuxostat 40 mg/day stably for ≥2 weeks during screening and run-in period,;
4. Meet the gout classification criteria formulated by the American College of Rheumatology (ACR) in 1977 or the joint gout classification criteria formulated by the American College of Rheumatology and the European League Against Rheumatism (ACR/EULAR) in 2015;
5. Body Mass Index (BMI) between 18 kg/m² and 35 kg/m².

Exclusion Criteria:

-

Subjects who meet any of the following conditions will be excluded:

1. General conditions:

1. Pregnant or lactating women;
2. Females of childbearing potential or males (except those whose partners are infertile) who refuse to use or use medically unapproved highly effective contraceptive measures within 6 months (for females) or 3 months (for males) from screening to the last dose of study medication;
3. Average daily alcohol intake exceeding 14 g for females (e.g., 145 mL of wine, 497 mL of beer, or 43 mL of low-alcohol liquor) or exceeding 28 g for males (e.g., 290 mL of wine, 994 mL of beer, or 86 mL of low-alcohol liquor) within 1 month before screening;
4. Drug abusers;
5. Subjects with poor compliance judged by investigators, which may affect the safety and efficacy evaluation of the study drug.

2. The following laboratory abnormalities within 4 weeks before randomization:

1. Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) and/or total bilirubin (TBIL) > 2 times the upper limit of normal (ULN);
2. Estimated glomerular filtration rate (eGFR) < 60 mL/(min×1.73m²) calculated by the Modification of Diet in Renal Disease (MDRD) formula based on serum creatinine level;
3. Glycated hemoglobin (HbA1c) ≥ 8%;
4. Active hepatitis B [positive hepatitis B surface antigen (HBsAg) and hepatitis B virus deoxyribonucleic acid (HBV-DNA) exceeding the normal range], or positive anti-hepatitis C virus (HCV) antibody, or positive human immunodeficiency virus (HIV) antibody, or positive syphilis antibody test;
5. White blood cell count < 3.0×10⁹/L, and/or hemoglobin < 90 g/L, and/or platelet count < 80×10⁹/L;
6. Prolonged QTcF interval confirmed by repeated 12-lead electrocardiogram (ECG) (QTcF > 450 ms).

3. History of or comorbidities with any of the following:

1. Hypersensitivity to SHR4640 or any component of SHR4640, or a history of intolerance or contraindication to febuxostat or citrate;
2. Secondary hyperuricemia caused by tumors, chronic kidney disease, hematological diseases, drugs, or other causes;
3. Other joint lesions that investigators believe may confuse gouty arthritis, such as rheumatoid arthritis, suppurative arthritis, traumatic arthritis, psoriatic arthritis, pseudogout, systemic lupus erythematosus, or joint lesions caused by chemotherapy, radiotherapy, chronic lead poisoning, acute obstructive nephropathy, etc.;
4. B-ultrasound suggesting or suspecting urinary calculi within 4 weeks before randomization;
5. Gout flare within 2 weeks before randomization;
6. History of active peptic ulcer within 1 year before screening and during the screening period, or active peptic ulcer at screening;
7. History of xanthinuria;
8. Suffering from malignant tumors, or a history of malignant tumors within 5 years before screening (except for treated non-melanoma skin cancers with no signs of recurrence and resected cervical intraepithelial neoplasia);
9. History of chronic or recurrent infections within 1 year before screening and during the screening period; or severe infections (including but not limited to hepatitis, sepsis, pneumonia, pyelonephritis, etc.) or infections leading to hospitalization within 3 months before screening and during the screening period; or infections treated with intravenous antibiotics within 2 weeks before randomization; or open draining wounds or ulcers at screening and during the screening period;
10. Subjects requiring systemic treatment with immunosuppressants;
11. Past or current moderate to severe congestive heart failure (New York Heart Association Class III or IV);
12. Myocardial infarction, unstable angina pectoris, percutaneous transluminal coronary angioplasty, coronary artery bypass grafting, cerebral infarction, cerebral hemorrhage, subarachnoid hemorrhage, transient ischemic attack, and other cardiovascular and cerebrovascular events leading to hospitalization within 1 year before screening and during the screening period;
13. Poorly controlled hypertension at screening and during the screening period [resting systolic blood pressure (SBP) ≥ 180 mmHg and/or diastolic blood pressure (DBP) ≥ 110 mmHg, confirmed by re-examination];
14. Complicated with other severe or poorly controlled diseases;
15. Major surgery performed within 3 months before screening and during the screening period, or failure to recover after surgery, or plan to undergo major surgery during the study;
16. Blood donation (or blood loss) with a volume ≥ 400 mL, or blood transfusion received within 3 months before screening and during the screening period;
17. Other conditions deemed inappropriate for participation in this study by investigators.

4. Use of any of the following drugs or participation in clinical trials:

1. Participation in any clinical trial of investigational drugs (including investigational vaccines) and use of investigational drugs within 3 months before screening or within 5 half-lives of the investigational drug (whichever is longer);
2. Participation in any clinical trial of medical devices within 3 months before screening (excluding subjects who failed screening);
3. Use of other urate-lowering drugs (allopurinol, probenecid, benzbromarone, dotinurad, recombinant urate oxidase) within 4 weeks before screening;
4. Use of drugs that interact with febuxostat (theophylline, azathioprine, mercaptopurine) within 4 weeks before screening;
5. Daily aspirin dosage exceeding 100 mg or unstable dosage within 4 weeks before screening;
6. Use of any diuretics within 2 weeks before randomization;
7. Use of angiotensin II receptor blockers (e.g., losartan), calcium channel blockers (e.g., amlodipine), fibrate lipid-lowering drugs (e.g., fenofibrate), statin lipid-lowering drugs (e.g., atorvastatin), clofibrate, acetohexamide, or sodium-glucose cotransporter 2 (SGLT2) inhibitors (e.g., empagliflozin) with unstable dosages within 2 weeks before randomization.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects with serum uric acid levels of ≤360 μmol/L at week 12 | at week 12

SECONDARY OUTCOMES:
Proportion of subjects with serum uric acid levels ≤300 μmol/L at week 12; | at week 12;
Proportion of subjects with serum uric acid levels ≤360 μmol/L at the last two test at week 12; | at week 12;
Proportion of subjects with serum uric acid levels ≤360 μmol/L at week 24; | at week 24;
Proportion of subjects with serum uric acid levels ≤300 μmol/L at week 24; | at week 24;
Proportion of subjects with serum uric acid levels ≤360 μmol/L at the last two test at week 24; | at week 24;
Percentage change in serum uric acid levels from baseline at each visit | within 24-week treatment period]
Change in serum uric acid levels from baseline at each visit | within 24-week treatment period
Proportion of subjects with serum uric acid levels ≤360 μmol/L at each visit | within 24-week treatment period

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided